CLINICAL TRIAL: NCT07026357
Title: Impact of 3D-planimetry on Optimized Therapeutic Assessment in Complex Benign Esophageal Stenosis; a Prospective Multi-center Study
Brief Title: Impact of 3D-planimetry on Optimized Therapeutic Assessment in Complex Benign Esophageal Stenosis
Acronym: INTENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Seufferlein (Other)
Collaborators: University Hospital Tuebingen (Other); University Hospital Augsburg (Other); University Hospital Munich (Other)
Responsible Party: Sponsor-Investigator, Thomas Seufferlein, Prof. Dr., University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UL001
Record Dates: First submitted 2022-06-07; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Benign Esophageal Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D-planimetric Measurement (Experimental): Esophageal stenosis is measured and endoscopic therapy is controlled by 3D-planimetry in addition to the conventional method (fluoroscopy, endoscopic examination)
  Interventions: Device: 3D-planimetric measurement; Radiation: Fluoroscopic control; Diagnostic Test: Endoscopic control
- Conventional Measurement (Active Comparator): Esophageal stenosis is measured and endoscopic therapy is controlled by fluoroscopy and endoscopic examination only
  Interventions: Radiation: Fluoroscopic control; Diagnostic Test: Endoscopic control

INTERVENTIONS:
Device: 3D-planimetric measurement — Esophageal stenosis is evaluated by 3D-planimetric measurement
  Arms: 3D-planimetric Measurement
Radiation: Fluoroscopic control — Fluoroscopic control of dilatation therapy
Diagnostic Test: Endoscopic control — Macroscopic endoscopic control of dilatation therapy

SUMMARY:
Esophageal stenosis has a high impact on patients quality of live and food intake affecting personal nutrition status and general health.

For benign strictures of the esophagus, endoscopic dilatation therapy is recommended by actual guidelines.

Since the extent of dilatation is currently directed by endoscopic view and fluoroscopic imaging, patients are exposed to radiation and the determination of the appropriate extent of dilatation is difficult.

Therefore, the aim of this study is to compare the effect of 3D-planimetric measurement with current fluoroscopic monitoring on the success of endoscopic esophageal dilatation therapy in patients with benign esophageal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic benign esophageal stenosis
* medical indication for endoscopic therapy
* written consent after detailed information

Exclusion Criteria:

* non-benign esophageal stenosis
* missing written consent
* trans-oral endoscopic access is not possible
* medical contraindication for endoscopic dilatation therapy
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Endoscopic therapy success | 3 months after intervention at endoscopic control examination
  Change in esophageal diameter [mm] and length of esophageal stricture [cm] after endoscopic therapy

SECONDARY OUTCOMES:
Length measurement of esophageal stenosis | during endoscopic intervention
  Length measurement of esophageal stenosis by different methods [cm]
Postinterventional esophageal diameter | directly after endoscopic intervention
  Postinterventional esophageal diameter [mm]
Hospitalization time after endoscopic dilatation therapy | within 3 months after study intervention
  Period of Hospitalization [days] after endoscopic dilatation therapy
Number of endoscopic interventions | within 3 months after study intervention
  Number of endoscopic interventions after study intervention
Number of hospitalizations due to complications | within 3 months after initial study intervention
  Hospitalization after study intervention [number of events, days] due to complications
Quality of life assessed by German Sydney Swallow Questionnaire | Baseline study intervention and 2 weeks after study intervention
  Quality of life according to the German Sydney Swallow Questionnaire (G-SWAL-QoL) questionnaire [17 questions, minimum 0 to maximum 1700 points; higher score indicates higher impairment considering swallowing]
Complication rate | during the procedure
  Peri-procedural complication rate
Duration of endoscopic examination | during the procedure
  Duration of endoscopic examination [minutes]
Sedation dose | during the procedure
  Dose of sedative medication [mg] during study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Walter, PhD, Principal Investigator — University Hospital Ulm
Locations (1):
- University Hospital Ulm, Clinic for Internal Medicine I, Ulm, Baden-Wuerttenberg, Germany

IPD SHARING:
Plan to Share IPD: No